CLINICAL TRIAL: NCT06846645
Title: Peripheral Blood Single Cell-type Expression Profile of Interferon-stimulated and Other Biomarker Genes for Triage of Febrile Patients
Brief Title: Host Response to Infection by Direct Analysis of Leukocyte Single Cell-type Gene Expression/transcript Abundance, Direct LS-TA. a Prospective Study Will Evaluate the Performance of Direct LS-TA in Triage Febrile Patients Into Major Categories of Infections: Viral, Bacterial or Active Tuberculosis.
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Nelson Tang, Principal Investigator, Chinese University of Hong Kong
Other Study IDs: Direct LS-TA prospective study
Record Dates: First submitted 2025-02-18; First posted 2025-02-26 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Single Cell Sequencing Technology; Gene Expression Profiling; Gene Expression; Infection; Viral Diseases; Bacterial Diseases; Active Tuberculosis; Host Defense Mechanisms; Host Microbial Interactions; Transcriptome
Keywords: host response; transcriptome; single cell-type gene expression; single cell RNA; triage; fever; febrile patient; Direct LS-TA
MeSH Terms: conditions — Infections; Virus Diseases; Bacterial Infections; Latent Tuberculosis; Fever

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood is collected into EDTA or citrate tubes. An aliquot of whole blood (WB) will be processed for RNA fixation by addition of Trizol solution and stored in -70C before total RNA extraction. Another aliquot of WB are separated into granulocytes and PBMC by the Ficoll gradient method. Granulocytes and a portion of PBMC will be fixed by Trizol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Bacterial infection group: A prospective sample of adult patients who later confirmed to have fever due to bacterial infection by positive culture results.
  Interventions: Other: No intervention
- Viral infection group: A prospective sample of adult patients who later confirmed to have fever due to viral infection by positive pathogen diagnostic results.
  Interventions: Other: No intervention
- Active tuberculosis group: A prospective sample of adult patients who later confirmed to have fever due to active tuberculosis by clinical diagnosis and/or positive pathogen results.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Patients will receive clinical treatment with no special intervention in this observational study. There is no difference in term of treatment of patients. It only involves one additional blood sampling early after admission.

SUMMARY:
Febrile illness is a common condition and it is crucial to have an early triage of patients according to various aetiologies to enable appropriate treatment. Currently, most screening/diagnostic tests target the detection of pathogens, while only a few assays aim to understand the host response, and they are mostly based on a measurement of serum proteins (e.g. CRP or procalcitonin).

Recently, blood transcriptome has been explored to differentiate bacterial and viral infections. However, gene expression in blood represents a composite score of gene expression of all the component cell-types present in the sample. Here, we propose to develop a rapid test that can determine gene expressions of a specified single cell type in peripheral blood (e.g., monocytes or granulocytes) as a host response biomarker to differentiate three major categories of infections that are bacterial, viral, and tuberculosis The assay is called Direct Leukocyte Single cell-type transcript abundance (TA) assay (DIRECT LS-TA) as it can directly determine the gene expression of a specified single cell-type among various other leukocyte populations directly in a peripheral blood sample. Such results signify the nature of host response according to 3 or more axes (Type I or Type II interferon signaling response or pro-inflammatory cytokine signaling) And it can be used to indicate the type of underlying infection (viral, bacterial, or active tuberculosis).

DETAILED DESCRIPTION:
DIRECT LS-TA is a ratio-based biomarker (RBB) for blood gene expression analysis which can be performed in commonly available equipments (e.g. qPCR or digital PCR machines). Using the ratio of TA of prior defined numerator gene and denominator gene, this RBB can quantify gene expression of the specified constitutional single cell-type (e.g. monocytes and granulocytes) inside a cell-mixture sample of Whole blood. DIRECT LS-TA was a method pioneered by the PI [Tang 2017, https://patents.google.com/patent/US9589099B2/]. And it has been developed for quantification of early B cell response after vaccination [DOI: 10.3390/genes12070971]. Recently, the method is used to develop host response biomarkers after infection to differentiate the type of pathogens (such as viral, bacterial or active tuberculosis). Numerator and denominator genes have been identified by using public gene expression datasets for monocytes and granulocytes. Diagnostic performance was good using these public data. Therefore, these RBBs will be applied in the prospective study to evaluate and compare their diagnostic (triage) performance of febrile patients into different pathogen etiologies.

Comparing to other methods to obtain single cell-type gene expression data, DIRECT LS-TA has many advantages The conventional (gold standard) approach is to quantify gene expression in a sample of purified single cell-type from peripheral blood but it is very labour intensive procedure. Recent single-cell RNA sequencing can also provide gene expression data for every individual cell in a sample, but it is slow and very costly. DIRECT LS-TA provides the unique technique to quantify single cell-type gene expression in blood samples without the need to isolate the targeted cell-type. It has been used to differentiate the type of host response in fever patients into 3 major axes (Type I or Type II interferon signaling response or pro-inflammatory cytokine signaling) which correspond to the nature of underlying infection aetiologies (viral infection, active tuberculosis and bacterial infection).

See preprint DOI: 10.1101/2025.01.27.634977. and patents in B cells : https://patents.google.com/patent/WO2022089426A1/ Monocytes: https://patents.google.com/patent/WO2023109365A1/ Granulocytes : https://patents.google.com/patent/GB202400180D0/

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with fever of acute onset which is defined by a raised body temperature.
* Patient should understand Chinese word to give informed consent.

Exclusion Criteria:

* Patients with a history of any immunodeficiency or immunocompromised condition. Patients received steriod or other immunotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with fever due to infections which are later clinically diagnosed as viral infection, bacterial infection or active tuberculosis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Viral host response Direct LS-TA in monocytes (Type I interferon response) | first collected sample within the first week after admission
  Direct LS-TA is a kind of RBB that can be readily quantified by qPCR or dPCR of a pair of genes, the RBB numerator gene and the RBB denominator gene. The biomarker is the ratio of the 2 genes. Single cell-type: Monocyte. RBB numerator gene: IFI27 or IFI44L. RBB denominator gene: PSAP, CTSS or CPVL.
  The various RBB (e.g. IFI27/PSAP and IFI44L/PSAP ratios) will be compared in terms of their sensitivity/specificity of diagnostic performance in the samples from infection groups. AUC of ROC analysis will be performed where appropriate.
Viral host response Direct LS-TA in granulocytes (Type I interferon response) | first collected sample within the first week after admission
  Direct LS-TA is a kind of RBB that can be readily quantified by qPCR or dPCR of a pair of genes, the RBB numerator gene and the RBB denominator gene. The biomarker is the ratio of the 2 genes. Single cell-type: Granulocyte. RBB numerator gene: RSAD2 or IFIT1.
  RBB denominator gene: SAT1 or SRGN. The various RBB will be compared in terms of their sensitivity/specificity of diagnostic performance in the infection groups. AUC of ROC analysis will be performed where appropriate.
Bacterial infection host response Direct LS-TA in monocytes (pro-inflammatory response) | first collected sample within the first week after admission
  Direct LS-TA is a kind of RBB that can be readily quantified by qPCR or digital PCR (dPCR) of a pair of genes, the RBB numerator gene and the RBB denominator gene. The biomarker is the ratio of the 2 genes. Single cell-type: Monocyte. RBB numerator gene: VNN1 or NLRC4. RBB denominator gene: PSAP, CTSS or CPVL. The various RBBs will be compared in terms of their sensitivity/specificity of diagnostic performance in the infection groups. AUC of ROC analysis will be performed where appropriate.
Bacterial infection host response Direct LS-TA in granulocytes (pro-inflammatory response) | first collected sample within the first week after admission
  Direct LS-TA is a kind of RBB that can be readily quantified by qPCR or dPCR of a pair of genes, the RBB numerator gene and the RBB denominator gene. The biomarker is the ratio of the 2 genes. Single cell-type: Granulocyte. RBB numerator gene: ALPL, ANXA3 or ARG1.
  RBB denominator gene: SAT1 or SRGN. The various RBB will be compared in terms of their sensitivity/specificity of diagnostic performance in the infection groups. AUC of ROC analysis will be performed where appropriate.
Active TB host response Direct LS-TA in monocytes (Type II interferon response) | first collected sample within the first week after admission
  Direct LS-TA is a kind of RBB that can be readily quantified by qPCR or dPCR of a pair of genes, the RBB numerator gene and the RBB denominator gene. The biomarker is the ratio of the 2 genes. Single cell-type: Monocyte.
  RBB numerator gene: WARS1, ATF3 or CALHM6. RBB denominator gene: PSAP, CTSS or CPVL. The various RBB will be compared in terms of their sensitivity/specificity of diagnostic performance in infection groups. AUC of ROC analysis will be performed where appropriate.
Active TB host response Direct LS-TA in granulocytes (Type II interferon response) | first collected sample within the first week after admission
  Direct LS-TA is a kind of RBB that can be readily quantified by qPCR or dPCR of a pair of genes, the RBB numerator gene and the RBB denominator gene. The biomarker is the ratio of the 2 genes. Single cell-type: granulocyte. RBB numerator gene: ANKRD22, BATF2, CD274, FCGR1A or ETV7.
  RBB denominator gene: SAT1 or SRGN. The various RBB will be compared in terms of their sensitivity/specificity of diagnostic performance in infection groups. AUC of ROC analysis will be performed where appropriate.

SECONDARY OUTCOMES:
DIRECT LS-TA results distribution and median of these DIRECT LS-TA RBB in infection groups | first collected sample within the first week after admission
  The statistical distribution of the biomarker and statistical comparison to the control range or comparison to control group median. The outcomes will be reported as p-values of the statistical tests.
Method evaluation to compare the performance of quantitative PCR and digital PCR | first collected sample within the first week after admission
  Evaluate the assay performance and precision of both TA quantification methods: quantitative PCR and digital PCR.
  Quantitative PCR results will be reported as delta-delta CT values. Digital PCR results will be reported as ratios of 2 counts. And then converted to multiple of mean/median in the control control (MoM) for comparison with delta-delta CT values.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Chemical Pathology, Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Descriptive statistics of results will be provided on a reasonable request.

REFERENCES:
- [Background] Huang D, Liu AYN, Leung KS, Tang NLS. Direct Measurement of B Lymphocyte Gene Expression Biomarkers in Peripheral Blood Transcriptomics Enables Early Prediction of Vaccine Seroconversion. Genes (Basel). 2021 Jun 25;12(7):971. doi: 10.3390/genes12070971. PMID 34202032
- [Background] Huang B, Huang J, Chiang NH, Chen Z, Lui G, Ling L, Kwan MYW, Wong JSC, Mak PQ, Ling JWH, Lam ICS, Ng RWY, Wang X, Gao R, Hui DS, Ma SL, Chan PKS, Tang NLS. Interferon response and profiling of interferon response genes in peripheral blood of vaccine-naive COVID-19 patients. Front Immunol. 2024 Jan 10;14:1315602. doi: 10.3389/fimmu.2023.1315602. eCollection 2023. PMID 38268924
- See also: Determination of gene expression levels of a cell type — https://patents.google.com/patent/US9589099B2/
- See also: Method for measuring gene expression of single cell subpopulation, related kit, and application — https://patents.google.com/patent/GB2629711A/en